CLINICAL TRIAL: NCT07202039
Title: Electronic Cigarettes as a Harm Reduction Strategy Among People With Opioid Use Disorder on Buprenorphine
Acronym: SWITCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Irene Pericot-Valverde, Assistant Professor, Clemson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2328661-1; K01DA062708 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Tobacco-flavored EC; Sweet-Cooling EC; Sweet Non-cooling EC
Keywords: Cigarette Smoking; Opioid use disorder; Burprenorphine; Electronic cigarettes; Switching; Flavors
MeSH Terms: conditions — Cigarette Smoking; Opioid-Related Disorders; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sweet-Cooling EC + Counseling (Experimental): Those randomized to the intervention group will be provided a free 12-week supply of sweet-cooling electronic cigarette (EC) liquid and five brief, individual counseling sessions, and asked to try to switch completely to EC.
  Interventions: Behavioral: Brief individual counseling sessions
- Sweet non-cooling EC + Counseling (Experimental): Those randomized to the intervention group will be provided a free 12-week supply of sweet non-cooling electronic cigarette (EC) liquid and five brief, individual counseling sessions, and asked to try to switch completely to EC.
  Interventions: Behavioral: Brief individual counseling sessions
- Tobacco-flavored EC + Counseling (Active Comparator): Those randomized to the intervention group will be provided a free 12-week supply of tobacco-flavored electronic cigarette (EC) liquid and five brief, individual counseling sessions, and asked to try to switch completely to EC.
  Interventions: Behavioral: Brief individual counseling sessions

INTERVENTIONS:
Behavioral: Brief individual counseling sessions — Five brief, individual counseling sessions will provide education, behavioral support, and motivational strategies to facilitate switching from combustible cigarette use to EC

SUMMARY:
This project aims to investigate the impact of e-cigarette flavors and usage patterns on achieving harm-reduction milestones in a sample of cigarette smokers with opioid use disorder who are taking buprenorphine

ELIGIBILITY:
Inclusion Criteria

* Age ≥21 years
* Smoke ≥5 CPD for ≥1 year
* Daily CC smoker
* Willing to switch to EC
* Exhaled CO ≥6 ppm
* Diagnosed with OUD
* Stable on bupropion treatment
* In good physical and mental health
* Able to use a smartphone
* Willing to participate in all study components
* Able to provide informed consent Exclusion Criteria
* Interested in quitting CC (contemplation stage of change)
* Use of EC on ≥4 of the past 30 days
* Use of other tobacco products (e.g., cigars, smokeless tobacco) on ≥9 days of the past 30 days
* Use of nicotine replacement therapy, smoking cessation medication, or a cessation attempt in the past 30 days
* Hypertension
* Medical condition that would contraindicate participation
* Meet DSM-V criteria for major depressive episode, psychotic episode, or manic episode
* Current suicidal ideation or suicide attempt in the past year
* Psychiatric hospitalization in the past year
* Contemplating pregnancy, currently pregnant, or breastfeeding
* Unable to speak and/or read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-10-27 (Estimated); Study Completion 2030-02-04 (Estimated)

PRIMARY OUTCOMES:
Change in cigarettes smoked per day | Baseline to week 12
  The average change in mean CPD on a 7-day TLFB assessment from baseline (week 0) to weeks 12

SECONDARY OUTCOMES:
Change in cigarettes smoked per day | Baseline to week 24
  The average change in mean CPD on a 7-day TLFB assessment from baseline (week 0) to week 24
Percentage of participants with a ≥50% reduction in CPD | Baseline to weeks 12 and 26
  The rate of participants achieving an average ≥50% reduction in CPD from baseline (week 0) to weeks 12 and 26, based on a 7-day TLFB
Switching | Weeks 12 and 24
  Proportion of participants reporting exclusive EC use and no CC use on a 7-day TLFB with CO <6 ppm.
Partial Switching | Weeks 12 and 24
  Proportion of participants reporting both EC and CC use on a 7-day TLFB with a ≥50% reduction in CPD.
7-Day CC Abstinence | Weeks 12 and 26
  Percentage of participants with biochemically verified 7-day abstinence (1 = abstinent, 0 = non-abstinent). Defined as self-reported no CC use on a 7-day TLFB with CO <6 ppm.
Change in carbon monoxide levels | Baselone to weeks 12 and 26
  Change in exhaled CO levels from baseline (week 0) to weeks 12 and 26 (continuous variable).

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction Medicine Center, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided